CLINICAL TRIAL: NCT01012791
Title: Does Zumba Improve Cognition in Healthy APOE e4 Carriers and Noncarriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Cynthia Stonnington, M.D., Mayo Clinic Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-000597
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Cognitive Impairment
Keywords: Zumba exercise; ApoE
MeSH Terms: conditions — Cognitive Dysfunction

ARMS (2):
- Zumba exercise group (Experimental)
  Interventions: Other: Zumba exercise
- Non-Zumba exercise group (No Intervention)

INTERVENTIONS:
Other: Zumba exercise — Subjects with do Zumba exercise for approximately 60 minutes twice a week for 6 months.
  Arms: Zumba exercise group

SUMMARY:
The main purpose of this study is to compare the effects on attention and memory functioning to participating in an aerobic and dance exercise called Zumba to educational program on exercise that encourages regular stretching and walking.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between the ages of 55-80 without cognitive complaints

Exclusion Criteria:

* History of significant health conditions

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To examine the feasibility of doing exercise intervention studies in presymptomatic, at risk individuals and determine the optimal outcome measure with minimal practice effect. | 6 months

SECONDARY OUTCOMES:
To examine whether forty 60 minute sessions of Zumba are associated with cognitive changes in healthy women between 55 and 80 years of age. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stonnington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States